CLINICAL TRIAL: NCT05611775
Title: Real-World Functional Activity in Adult Spinal Deformity Surgery
Brief Title: Adult Spinal Deformity Surgery Real-World Functional Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin D. Elder, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-007211
Record Dates: First submitted 2022-11-01; First posted 2022-11-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Thoracolumbar Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Activity Monitor Assessment (Other): Subjects will be assessed in the Motion Analysis Laboratory at Mayo Clinic Rochester and have activity monitored in the free-living environment.
  Interventions: Device: Triaxial accelerometer

INTERVENTIONS:
Device: Triaxial accelerometer — Monitors placed on the waist, thigh, and bilateral ankles. Accelerometry will measure patients' physical activities in the free-living environment for 4 consecutive days. The patients will wear the monitor during waking hours and remove it during sleeping, showering, and swimming time.

SUMMARY:
The purpose of this study is to measure functional activity and stability in spinal deformity patients utilizing motion analysis testing and accelerometers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of degenerative thoracolumbar deformity
* Deformity correction surgery scheduled with either Dr. Elder or Dr. Fogelson, minimum 4-level fusion with fixation to the pelvis.

Exclusion Criteria:

° Unable to return to Mayo Clinic for follow-up evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Motion Analysis Lab - Change in function | Baseline, 6-12 weeks post-surgery, 1 year
  Spatiotemporal measures including velocity, step/stride length, step width, single/double support times, and R/L temporal symmetriesm will be used to measure function.
Motion Analysis Lab - Change in gait | Baseline, 6-12 weeks post-surgery, 1 year
  Gait will be measured by segmental and joint range of motion, peak kinetics during walking, and changes in deviation from normal bands using sensory processing measures.
Motion Analysis Lab - Change in trunk stability | Baseline, 6-12 weeks post-surgery, 1 year
  Trunk stability will be measured by EMG frequency content and activation pattern during gait and postural sway.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Elder, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No